CLINICAL TRIAL: NCT00664300
Title: Facial Expression Recognition of Emotion and Categorization of Emotional Words in Gilles de la Tourette's Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pr Jalenques, CHU Clermont-Ferrand
Other Study IDs: CHU-0032; RBHP 2007 Jalenques
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Gilles de la Tourette's Syndrome
Keywords: Gilles de la Tourette's syndrome; Facial expression recognition of emotion; Frequency levels; Automatic and voluntary information treatment; Patient with Gilles de la Tourette's syndrome
MeSH Terms: conditions — Tourette Syndrome

GROUPS / COHORTS (1):
- 2: One group with Gilles de la Tourette's Syndrome One group with healthy paired volunteers
  Interventions: Behavioral: Facial expression recognition of emotion

INTERVENTIONS:
Behavioral: Facial expression recognition of emotion — Facial expression recognition test Lexical decision test

SUMMARY:
Gilles de la Tourette's syndrome is a childhood onset inherited neuropsychiatric disorder characterised by the presence of both multiple motor tics and one or more vocal tics (noises), with psychiatric and/or behaviour disorders (such as obsessive compulsive behaviour…).

This disease is associated with an dopamine system imbalance which could be responsible of a specific trouble in the recognition in some facial expression. This has been already shown in Gilles de la Tourette patients with obsessive compulsive behaviour.

We hypothesise that patients with Gilles de la Tourette's syndrome present a dysfunction of voluntary and automatic treatment of emotional information.

The main purpose of this study is to show if patients with Gilles de la Tourette's syndrome present a lack of specific facial expression recognition of emotion and determinate more precisely if this alteration involves the cortical way (high frequency way) or the under cortical way (low frequency way).

DETAILED DESCRIPTION:
20 patients with Gilles de la Tourette's syndrome compared to 20 healthy paired volunteers.

Study progress (patients):

Inclusion visit :

Psychiatric evaluation Psychological evaluation

Ophthalmic visit

Protocol :

Facial expression recognition test Lexical decision test

Study progress (healthy volunteers):

Psychiatric evaluation Ophthalmic visit Facial expression recognition test Lexical decision test

ELIGIBILITY:
Inclusion Criteria:

* Age : >18 years
* Patient with a Gilles de la Tourette 's syndrome such as defined in the DSMIV
* Stability of treatment >1 month
* Mini Mental State > 26
* Affiliation to social security
* Agreement of patients

Exclusion Criteria:

* Patients with cognitive disorders, dementia, mental retardation…
* Patients with serious neurological pathologies
* Patients with a vision contrast altered.
* Patients who do not understand the words associated with an emotion
* Pregnant women
* Person who participate to an other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with Gilles de la Tourette's Syndrome and 30 healthy paired volunteers (control group)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Facial expression recognition test | % of exact responses

SECONDARY OUTCOMES:
Lexical decision test | The time to respond

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Jalenques, PUPH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France